CLINICAL TRIAL: NCT01816503
Title: High-dose Fentanyl Matrix Application for Cancer Pain: Multicenter, Prospective, Observational Study
Brief Title: Fentanyl Matrix Application for Cancer Pain: Multicenter, Prospective, Observational Study
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015778; FENPAI4084 (Other: Janssen Korea, Ltd., Korea); FEN-KOR-5027 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: Pain; Cancer pain; Fentanyl; Fentanyl matrix; Opioid analgesic
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fentanyl matrix
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. The minimum initial dose will be fentanyl matrix 75 micrograms/h and the investigator can adjust the dosage according to the degree of the patients' pain control during the 9 days of the study period. Fentanyl matrix is a transdermal patch that is applied on the patient's skin.

SUMMARY:
The purpose of this study is to show the clinical usefulness of fentanyl matrix by measuring satisfaction with pain treatment after administering fentanyl matrix in patients whose pain was not controlled sufficiently with the previous analgesic use in real practice at the investigator's discretion.

DETAILED DESCRIPTION:
This is a multi-center, open-label (all people know the identity of the intervention), prospective (the patients are identified and then followed forward in time for the outcome of the study) observational study. The study population comprises patients who are admitted to a study center during the study period and are receiving a strong oral long-acting opioid analgesic but deemed to control pain insufficiently. Since this study is an observational study conducted in real practice, a dose of fentanyl matrix should be adjusted depending on an individual patient's response at the investigator's discretion. However, for the patients whose pain is not sufficiently controlled despite administration of strong long-acting opioid analgesics, the minimum initial dose will be fentanyl matrix 75 micrograms/h and the investigator can adjust dosage according to the degree of the patients' pain control during the 9 days of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of cancer pain which requires administration of long-acting opioid analgesics
* Patients whose pain is not sufficiently controlled despite administration of strong long-acting opioid analgesics
* Patients who are deemed to need an initial minimum dose of fentanyl matrix 75 micrograms/h
* Patients who signed the informed consent form

Exclusion Criteria:

* Patients with a history of or current drug or alcohol abuse
* Childbearing women who are pregnant or likely to be pregnant during the study period and men who are neither infertile nor willing to refrain from sexual relations but whose partner does not conduct an effective contraception
* Patients who are unable to use a transdermal system due to skin disease
* Patients with history of hypersensitivity to opioid analgesics
* Patients who are not eligible for the study participation based on warnings, precautions and contraindications in the package insert of the study drug at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to a study center during the study period and are receiving a strong oral long-acting opioid analgesic but deemed to control pain insufficiently.
Sampling Method: Non-Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who are very satisfied or satisfied with the pain treatment after the study drug administration | Day 10
  The overall satisfaction is measured by a 5-point scale. Patients' answers are rated as: "very satisfied", "satisfied", "fair", "dissatisfied", or "very dissatisfied".

SECONDARY OUTCOMES:
The change from baseline in pain intensity | Baseline, up to Day 10
  The mean pain intensity the patient experienced over the last 24 hours will be measured through Numeric Rating Scale (NRS); 0 = no pain, 10 = worst pain imaginable.
The change from baseline in Karnofsky Performance Status Scale | Baseline, Day 10
  Karnofsky Performance Status Rating Scale is a tool to assess cancer patients' physical functioning. Scores range from 0 per cent (dead) to 100 per cent (normal, no complaints, no evidence of disease) in a unit of 10 per cent to indicate a level of overall daily activity performance status.
Sleep disturbance caused by the number of awakening caused by pain the patient experienced over the last night | 10 days
  Patients indicate in a Numeric Rating Scale (NRS) the number of awakening from sleep due to pain in the previous night: not awakened, once, twice, more than 3 times, or could not sleep.
Sleep disturbance caused by pain the patient experienced over the last 24 hours | 10 days
  Patients indicate in a Numeric Rating Scale (NRS) the sleep disturbance caused by pain experienced over the last 24 hours, where 0= not disturbing at all, and 10= very disturbing.
The change from baseline in Clinical Global Impression - Improvement (CGI-I) | Baseline, Day 10
  CGI-I measures the overall improvement of the patient's condition compared to baseline, as follows; 1 = Improved very much, 2 = Improved a lot, 3 = Improved a little, 4 = No change, 5 = Aggravated a little, 6= Aggravated a lot, 7= Aggravated very much.
Patient's Global Assessment | Day 10
  This tool assesses how effective the study drug has been in pain treatment during the study period. The patient will assess the effectiveness from his/her viewpoint at visit 10 on a 5-point rating scale; 1 = not effective, 2 = fair, 3 = effective, 4 = very effective, 5 = very much effective.
Investigator's Global Assessment | Day 10
  This tool assesses how effective the study drug has been during the study period. The investigator will assess the effectiveness from his/her viewpoint at Visit 10 on a 5-point rating scale; 1 = not effective, 2 = fair, 3 = effective, 4 = very effective, 5 = very much effective.
Dose of fentanyl matrix | 9 days
  The dose of fentanyl matrix used throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea